CLINICAL TRIAL: NCT05819424
Title: EpiCor Clinical Study on Rapid Immune Modulating Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cargill (Industry)
Collaborators: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 004-044
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Immune Surveillance

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, randomized, double-blind, cross-over design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo intervention first and Active intervention one week later (Experimental): Participants will be consuming a placebo on a clinic day at least one week prior to a clinic day where they will consume the active intervention.
  Interventions: Dietary Supplement: Yeast Fermentate (EpiCor)
- Active intervention first and Placebo intervention one week later (Experimental): Participants will be consuming active intervention on a clinic day at least 1 week prior to a clinic day where they will consume the placebo.
  Interventions: Dietary Supplement: Yeast Fermentate (EpiCor)

INTERVENTIONS:
Dietary Supplement: Yeast Fermentate (EpiCor) — Dietary Supplement: Yeast Fermentate (EpiCor): Postbiotic whole food fermentate made using yeast. Composed of proteins, polyphenols, vitamins, minerals, amino acids, polysaccharides, fibre, and other nutrients.
  Placebo: Substance with no therapeutic value to facilitate blinding

SUMMARY:
Clinical verification study evaluating the effects of a nutraceutical product. This study involves thirty participants composed of healthy adults, who will be taking either a placebo or nutraceutical supplement at different times. Testing for immune status, cytokine levels, and immune responsiveness will be conducted to determine the acute impact of the nutraceutical on immune function compared to a placebo.

DETAILED DESCRIPTION:
Clinical study comparing the acute immune effect of a nutraceutical product and a placebo. The nutraceutical supplement is a postbiotic whole food fermentate produced using yeast.

30 subjects will participate in a placebo-controlled, double-blind, randomized, cross-over design, wherein they will be taking a placebo, or nutraceutical product, each separated by a 1-week washout period to evaluate effects within 3 hours of consumption.

Blood samples will be taken 1 hour after participants arrive, then the dose is administered. Samples are taken 1 hour, 2 hours, and 3 hours following administration.

A series of immune panels will be used to determine the acute impacts on immune surveillance, immune cell activation status, and cytokine profiles. Ex vivo immune challenges will be used to determine the direct impacts on immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of any gender
* BMI between 18 and 30 (inclusive)
* Veins easy to see in one or both arms (to allow for multiple blood draws)
* Willing to comply with a 24-h wash-out period for vitamins and nutritional supplements
* Willing to comply with study procedures including: maintaining a consistent diet and lifestyle routine throughout the study; consistent habit of bland breakfasts on days of clinic visits; abstaining from exercising and nutritional supplements on the morning of the study visit; abstaining from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit; abstaining from music, candy, bum, computer/cell phone use, during clinic visits.

Exclusion Criteria:

* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery not a problem, including previous removal of appendix and gall bladder)
* Currently in intensive athletic training (such as marathon runners)
* Currently taking antidepressant or tranquilizing medications
* Taking anti-inflammatory medications on a daily basis
* Currently experiencing intense stressful events/life changes that could negatively affect compliance
* Anything that the investigator judges may put the subject at risk or may unduly influence any of the results of the study
* An unusual sleep routine (examples: working nightshift, irregular routine with frequent late nights)
* Unwilling to maintain a constant intake of supplements over the duration of the study
* Anxiety about having blood drawn
* People of childbearing potential: pregnant, nursing, or trying to become pregnant
* Known food allergies related to ingredients in active test product or placebo

Prescription medication will be evaluated on case-by-case basis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Immune Surveillance | At 1, 2, and 3 hours
  Observation of changes in immune cell trafficking and status of immune cell alertness, i.e., the changes in immune cell populations and activation following administration

SECONDARY OUTCOMES:
Immune Communication | At 1, 2, and 3 hours
  Serum cytokine levels as assessed by changes in cytokine levels individually versus placebo

OTHER OUTCOMES:
Immune Responsiveness | At 1, 2, and 3 hours
  Ex vivo immune challenges, observing the capabilities of anti-bacterial and anti-viral defenses. Additionally, mucosal immune protection as determined by salivary IgA, defensins, and transferrin changes.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Jensen, PhD, Principal Investigator — NIS Labs
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No